CLINICAL TRIAL: NCT00294580
Title: Comparison of Two Strategies for Control of Malaria Within A Primary Health Care Programme in the Gambia
Brief Title: Early Childhood Malaria Prevention With Maloprim in The Gambia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council Unit, The Gambia (Other); Government of the Gambia (Unknown); London School of Hygiene and Tropical Medicine (Other); Partnership for Child Development (Unknown); Wellcome Trust (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: SCC-795-835
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Malaria
Keywords: Malaria; Cognition; Prevention & control; Anemia; Chemoprophylaxis; Mortality; Children; Randomized controlled trial; Education; Long-term effects; The Gambia; Africa, West
MeSH Terms: conditions — Malaria; Anemia | interventions — Maloprim

INTERVENTIONS:
Drug: Maloprim

SUMMARY:
A trial was conducted in the 1980s to compare two strategies for control of malaria in young children aged 3-59 months: treatment with chloroquine versus treatment combined with fortnightly chemoprophylaxis with Maloprim. The impact on mortality and morbidity was assessed at the time, and their cognitive abilities and educational outcomes were assess 14 years later in 2001. The hypothesis was that the chemoprophylaxis would reduce morbidity and mortality and would improve cognitive abilities and educational outcomes in the long term

DETAILED DESCRIPTION:
Two drug strategies for the control of malaria in children aged 3-59 months have been compared in a rural area of The Gambia - treatment of presumptive episodes of clinical malaria with chloroquine by village health workers, and treatment combined with fortnightly chemoprophylaxis (pyrimethamine/dapsone) which was also given by village health workers. Treatment alone did not have any significant effect on mortality or morbidity from malaria. In contrast, treatment and chemoprophylaxis reduced overall mortality in children aged 1-4 years, mortality from probable malaria, and episodes of fever associated with malaria parasitaemia. A high level of compliance with chemoprophylaxis was obtained and no harmful consequences of chemoprophylaxis were observed. Chemoprophylaxis was offered to all children at the end of the trial.

14 years after the end of the trial, participants cognitive abilities and educational attainment were assessed. Associations have been found between malaria infection and poor cognitive ability but causality has not yet been demonstrated through preventative trials and the long-term impact of malaria has not been investigated. 1190 children who had participated in the original trial for at least one year were targetted for follow-up. 579 were traced. Those who had received chemoprophylaxis attended school for 0.52 years more than the placebo group (p=.069). There was no overall effect on cognitive abilities but there was a significant treatment effect for cohorts that had not received chemoprophylaxis at the end of the trial or who had received less than one year of post-trial prophylaxis

ELIGIBILITY:
Inclusion Criteria:

* For original trial: Children aged 3-59 months present in participating villages
* For follow-up: Children who were in original trial for at least 1 year.

Exclusion Criteria:

* For original trial: None
* For follow-up: Children with mental or physical disabilities who were unable to do cognitive tests

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2253
Dates: Start 1982-04; Study Completion 2001-09

PRIMARY OUTCOMES:
Mortality
Episodes of Fever Associated with Malaria Parasitaemia
Cognitive Abilities in late adolescence
Educational Attainment (Years spent at school)

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Greenwood, MD, Principal Investigator — London School of Hygiene and Tropical Medicine; Matthew CH Jukes, DPhil, Principal Investigator — Imperial College London
Locations (1):
- Medical Research Council Field Station, Farafenni, Central River Division, The Gambia

REFERENCES:
- [Result] Greenwood BM, Greenwood AM, Bradley AK, Snow RW, Byass P, Hayes RJ, N'Jie AB. Comparison of two strategies for control of malaria within a primary health care programme in the Gambia. Lancet. 1988 May 21;1(8595):1121-7. doi: 10.1016/s0140-6736(88)91949-6. PMID 2896957
- [Result] Menon A, Snow RW, Byass P, Greenwood BM, Hayes RJ, N'Jie AB. Sustained protection against mortality and morbidity from malaria in rural Gambian children by chemoprophylaxis given by village health workers. Trans R Soc Trop Med Hyg. 1990 Nov-Dec;84(6):768-72. doi: 10.1016/0035-9203(90)90071-l. PMID 2096501
- [Result] Greenwood BM, David PH, Otoo-Forbes LN, Allen SJ, Alonso PL, Armstrong Schellenberg JR, Byass P, Hurwitz M, Menon A, Snow RW. Mortality and morbidity from malaria after stopping malaria chemoprophylaxis. Trans R Soc Trop Med Hyg. 1995 Nov-Dec;89(6):629-33. doi: 10.1016/0035-9203(95)90419-0. PMID 8594677